CLINICAL TRIAL: NCT05548569
Title: Relationship Between Vascular Endothelial Dysfunction and Beat-to-beat Blood Pressure Variability in Patients With Obstructive Sleep Apnea Syndrome
Brief Title: Relationship Between Vascular Endothelial Dysfunction and Beat-to-beat Blood Pressure Variability in Patients With OSAS
Status: Recruiting | Type: Observational
Sponsor: Huai'an No.1 People's Hospital (Other)
Responsible Party: Principal Investigator, Xu J, Deputy director, Huai'an No.1 People's Hospital
Other Study IDs: Huaian1PH3
Record Dates: First submitted 2022-09-16; First posted 2022-09-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-02

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Obstructive sleep apnea,endothelial dysfunction
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
It is thought that intermittent hypoxia, poor tissue oxygenation, and perfusion in OSA can lead to eNOS uncoupling. Uncoupled eNOS can reduce nitric oxide (NO), which will result in an imbalance of contraction and diastole. Furthermore, OSA may increase beat-to-to BPV via the characteristic acute blood pressure peaks that follow the end of obstructive apnoeas. Therefore, the aim is to discuss the relationship between vascular endothelial dysfunction and beat-to-beat blood pressure variability in patients with OSAS (Obstructive sleep apnea syndrome).

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is characterized by recurrent airway collapse that causes chronic intermittent hypoxia(CIH). OSA is associated with systemic inflammation and oxidative stress resulting in endothelial dysfunction and cardiovascular disease (CVD). Under physiological conditions, eNOS is activated by shear stress and Ach. L-arginine and O2 are catalyzed by BH4, FMN, FAD, NADPH, and eNOS to produce nitric oxide (NO)， which has an important vasodilating effect， and L-citrulline. During the episode of OSA, intermittent hypoxia leads to oxidative stress resulting in the production of superoxide anions. The reaction between O2- and NO occurs rapidly, resulting in ONOO-. ONOO- and H2O2 oxidize BH4 to dihydrobiotrexate (BH2), which is a competitive inhibitor with BH4, thus limiting the availability of eNOS substrates and preventing NO production, resulting in an imbalance between contraction and diastolic. It has been documented that beat-to-beat blood pressure variability in OSAS patients is much higher than that in healthy adults. In some patients, intermittent hypoxia was observed with the episode of OSA, and blood pressure fluctuated with the episode of hypoxia. However, this was not found in the other patients, whose blood pressure did not change significantly during the hypoxia episode. Therefore, the investigators considered that the endothelial function of patients with high sensitivity to hypoxia was healthy or in the early stage, while the endothelial function of those patients with low sensitivity to hypoxia was at a relatively high level of impairment. Endothelial dysfunction can be measured indirectly by brachial artery flow-mediated dilation (FMD), beat-to-beat blood pressure variability can be measured by Polysomnography (PSG), and biological examinations can be performed by blood sampling. Thus, the purpose is to explore the specific relationship between OSAS beat-to-beat blood pressure variability and endothelial dysfunction.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old;
2. Moderate to severe OSA(AHI≥15 times/hour);
3. Hypertension (systolic blood pressure ≥140mmHg and/or diastolic blood pressure ≥90mmHg);

Exclusion Criteria:

1. Malignant tumor, severe arrhythmia and heart disease, moderate and severe renal dysfunction, peripheral vascular disease, diabetes
2. Systolic blood pressure ≤140mmHg and diastolic blood pressure ≤90mmHg
3. Vigorous exercise 24 hours before the experiment;
4. Vasoactive drugs (ACEI, ARB, CCB, β blockers, nitrates) were used 48 hours before the experiment;
5. Smoking, drinking and consuming caffeinated beverages 12 hours before the experiment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatient snoring patients will have PSG, and patients aged 18 years and older will be included in the study.Inclusion Criteria:1. Moderate to severe OSA(AHI≥15 times/hour);2. Hypertension (systolic blood pressure ≥140mmHg and/or diastolic blood pressure ≥90mmHg);Exclusion Criteria:1.Malignant tumor, severe arrhythmia and heart disease, moderate and severe renal dysfunction, peripheral vascular disease, diabetes 2.Systolic blood pressure ≤140mmHg and diastolic blood pressure ≤90mmHg 3.Vigorous exercise 24 hours before the experiment; 4.Vasoactive drugs (ACEI, ARB, CCB, β blockers, nitrates) were used 48 hours before the experiment;
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Relationship Between Vascular Endothelial Dysfunction and Beat-to-beat Blood Pressure Variability in Patients With OSAS | 2022.04.01-2023.04.01
  the endothelial dysfucntion patients with OSAS have more sever blood pressure variability

CONTACTS AND LOCATIONS:
Locations (1):
- Jing Xu, Huai'an, Jiangsu, China

REFERENCES:
- [Background] Pal A, Martinez F, Aguila AP, Akey MA, Chatterjee R, Conserman MGE, Aysola RS, Henderson LA, Macey PM. Beat-to-beat blood pressure variability in patients with obstructive sleep apnea. J Clin Sleep Med. 2021 Mar 1;17(3):381-392. doi: 10.5664/jcsm.8866. PMID 33089774
- [Background] Dissanayake HU, Sutherland K, Phillips CL, Grunstein RR, Mihailidou AS, Cistulli PA. Comparative effects of CPAP and mandibular advancement splint therapy on blood pressure variability in moderate to severe obstructive sleep apnoea. Sleep Med. 2021 Apr;80:294-300. doi: 10.1016/j.sleep.2021.01.059. Epub 2021 Feb 3. PMID 33610954
- [Background] Sun Y, Liu F, Zhang Y, Lu Y, Su Z, Ji H, Cheng Y, Song W, Hidru TH, Yang X, Jiang Y. The relationship of endothelial function and arterial stiffness with subclinical target organ damage in essential hypertension. J Clin Hypertens (Greenwich). 2022 Apr;24(4):418-429. doi: 10.1111/jch.14447. Epub 2022 Mar 3. PMID 35238151
- [Background] Tatasciore A, Di Nicola M, Tommasi R, Santarelli F, Palombo C, Parati G, De Caterina R. From short-term blood pressure variability to atherosclerosis: Relative roles of vascular stiffness and endothelial dysfunction. J Clin Hypertens (Greenwich). 2020 Jul;22(7):1218-1227. doi: 10.1111/jch.13871. Epub 2020 Jul 8. PMID 32639102
- [Background] Genovesi S, Giussani M, Orlando A, Lieti G, Viazzi F, Parati G. Relationship between endothelin and nitric oxide pathways in the onset and maintenance of hypertension in children and adolescents. Pediatr Nephrol. 2022 Mar;37(3):537-545. doi: 10.1007/s00467-021-05144-2. Epub 2021 Jun 3. PMID 34085102